CLINICAL TRIAL: NCT01550783
Title: Cytology vs. at Home HPV Screening for Detection of CIN 2,3,CIS
Brief Title: Home-Based or Clinic-Based Human Papillomavirus (HPV) Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 7489; NCI-2013-00745 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7489 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA157469 (NIH)
Record Dates: First submitted 2012-02-17; First posted 2012-03-12 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2018-04

CONDITIONS: Atypical Squamous Cell of Undetermined Significance; Cervical Carcinoma; Cervical Intraepithelial Neoplasia Grade 2/3; Health Status Unknown; Human Papillomavirus Infection; Low Grade Cervical Squamous Intraepithelial Neoplasia; Stage 0 Cervical Cancer
Keywords: Cervical cancer; Atypical squamous cells of undetermined significance; Stage 0 cervical cancer; Cervical intraepithelial neoplasia grade 1; Cervical; intraepithelial neoplasia grade 2; Cervical intraepithelial neoplasia grade 3; Human papillomavirus; HPV
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; Uterine Cervical Dysplasia; Atypical Squamous Cells of the Cervix | interventions — Vaginal Smears; High-Throughput Screening Assays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (home-based HPV screening) (Experimental): Participants collect 2 vaginal specimens using polyester swabs that are then placed in a specimen tube. Specimens are then submitted to the Harborview Medical Center clinical pathology lab. Participants with a positive HPV test result will have a Pap test. Participants with an abnormal Pap test will undergo standard of care as in Group II.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Questionnaire Administration; Procedure: Screening Method
- Group II (clinic-based standard of care screening) (Experimental): Participants undergo standard of care cervical cancer screening and follow-up. That is, participants undergo Pap testing. Participants with an abnormal Pap test undergo HPV testing, colposcopy, cervical biopsy and/or ECC. Participants with cervical biopsies showing precancerous changes are offered to undergo LEEP or are referred to appropriate care.
  Interventions: Other: Cervical Papanicolaou Test; Other: Questionnaire Administration; Procedure: Screening Method

INTERVENTIONS:
Other: Cervical Papanicolaou Test — Undergo standard of care Pap test screening
  Other Names: Cervical Pap Test
  Arms: Group II (clinic-based standard of care screening)
Other: Cytology Specimen Collection Procedure — Undergo home-based HPV screening
  Other Names: Cytologic Sampling
  Arms: Group I (home-based HPV screening)
Other: Questionnaire Administration — Ancillary studies
Procedure: Screening Method — Undergo standard of care Pap test screening
  Arms: Group II (clinic-based standard of care screening)
Procedure: Screening Method — Undergo home-based HPV screening
  Arms: Group I (home-based HPV screening)

SUMMARY:
This randomized clinical trial studies home-based HPV or clinic-based Pap screening for cervical cancer. It is not yet known whether home-based screening is more effective, cost-effective, and/or acceptable than clinic-based screening for cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the sensitivity and specificity for cervical intraepithelial neoplasia (CIN) of two screening approaches:

* Novel approach: every 3 years high risk-human papillomavirus (HR-HPV) testing of (at home) self-collected samples with in-clinic cytology of HR-HPV positive women and referral to colposcopy of women with cytology > atypical squamous cells of uncertain significance (ASCUS); repeat HPV testing of HR-HPV positive but cytology negative women at one year;
* Currently recommended approach: for women < 30: every 3 years in-clinic cytology screening, with HPV based triage of women with ASCUS and referral to colposcopy of all women with squamous intraepithelial lesion (SIL) and/or HPV+ ASCUS; for women 30+, screening by Papanicolaou (Pap) and HPV, every 2-3 year (depending on previous history) with referral to colposcopy of those who are HPV 16/18+ or with cytology > ASCUS; retesting of those who are positive for other HR-HPV at one year.

II. Compare these two approaches with respect to overall cost-effectiveness and acceptability.

III. Determine the performance and cost-effectiveness of each approach in vaccinated and unvaccinated women < 30.

OUTLINE: Participants are randomized to 1 of 2 arms.

GROUP I (home-based HPV screening): Participants collect 2 vaginal specimens using polyester swabs. Participants with a positive HPV test result will have a Pap test. Participants with an abnormal Pap test will undergo standard of care as in Group II.

GROUP II (clinic-based standard of care screening): Participants undergo Pap testing. Participants with a positive Pap test undergo standard of care, including colposcopy, HPV testing, cervical biopsy and/or endocervical curettage (ECC). Participants with cervical biopsies showing precancerous changes requiring treatment may undergo loop electrosurgical excision procedure (LEEP) or are referred to appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent in English

Exclusion Criteria:

* Have had hysterectomy
* Currently pregnant
* Received treatment of cervical dysplasia with LEEP, cone biopsy, laser procedure or cryotherapy within THREE years
* Received colposcopy of cervix within TWO years
* Received Pap test within ONE year
* Immunocompromised (positive human immunodeficiency virus [HIV] test, transplant recipient, received chemotherapy for cancer, or taking immunosuppressant drugs)
* Decisionally impaired adults requiring a legally authorized representative

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1335 (Actual)
Dates: Start 2012-03; Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness in the novel approach in vaccinated and unvaccinated women less than 30 years old | Up to 4 years
Cost-effectiveness in the standard approach in vaccinated and unvaccinated women less than 30 years old | Up to 4 years
Overall cost-effectiveness and acceptability | Up to 4 years
  The results from the trial (sensitivity, specificity, and costs) will be used in conjunction with a Markov model to determine cost per LY and cost per QALY. Model outcomes (per 100,000 screened) will include the expected numbers of false-positive test results, colposcopies, cases of CIN 1+, cases of cancer, cancer deaths, life expectancy and quality adjusted life-expectancy. Strategies will be compared using incremental cost-effectiveness ratios. Costs and outcomes will be discounted at 3% annually. One, 2-way and probabilistic sensitivity analyses conducted for all inputs to the models.
Sensitivity and specificity for CIN 1+ of currently recommended in-clinic cytology screening | Up to 4 years
  An intention-to-treat analysis, based upon the initial randomization, will be performed to evaluate differences between study arms (screening strategies). Estimates of sensitivity and specificity for detection of CIN 1+ will be calculated for the two screening strategies using standard methodologies.
Sensitivity and specificity for CIN 1+ of novel home-based testing | Up to 4 years
  An intention-to-treat analysis, based upon the initial randomization, will be performed to evaluate differences between study arms (screening strategies). Estimates of sensitivity and specificity for detection of CIN 1+ will be calculated for the two screening strategies using standard methodologies.
Sensitivity and specificity of the novel approach in vaccinated women less than 30 years old | Up to 4 years
  Estimates of sensitivity and specificity for detection of CIN 1+ will be calculated for the two screening strategies and the rate of disease in the 10% sample of test negative subjects in each arm will be extrapolated to the entire study group of test negative subjects in that arm when sensitivity and specificity estimates are calculated. Threshold analyses will also be conducted to identify the range for the cost of the home-based test due to inherent uncertainty
Sensitivity and specificity of the standard approach in vaccinated women less than 30 years old | Up to 4 years
  Estimates of sensitivity and specificity for detection of CIN 1 will be calculated for the two screening strategies and the rate of disease in the 10% sample of test negative subjects in each arm will be extrapolated to the entire study group of test negative subjects in that arm when sensitivity and specificity estimates are calculated. Threshold analyses will also be conducted to identify the range for the cost of the home-based test due to inherent uncertainty

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Kiviat, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Feder MA, Kulasingam SL, Kiviat NB, Mao C, Nelson EJ, Winer RL, Whitham HK, Lin J, Hawes SE. Correlates of Human Papillomavirus Vaccination and Association with HPV-16 and HPV-18 DNA Detection in Young Women. J Womens Health (Larchmt). 2019 Oct;28(10):1428-1435. doi: 10.1089/jwh.2018.7340. Epub 2019 Jul 2. PMID 31264912
- [Derived] Mao C, Kulasingam SL, Whitham HK, Hawes SE, Lin J, Kiviat NB. Clinician and Patient Acceptability of Self-Collected Human Papillomavirus Testing for Cervical Cancer Screening. J Womens Health (Larchmt). 2017 Jun;26(6):609-615. doi: 10.1089/jwh.2016.5965. Epub 2017 Mar 23. PMID 28332888